CLINICAL TRIAL: NCT00034372
Title: Multicenter Clinical Trial of Intravenous OvaRex MAb-B43.13 as Post-Chemotherapy Consolidation for Ovarian Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: closed by sponser
Sponsor: Unither Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OVA-Gy-15
Record Dates: First submitted 2002-04-26; First posted 2002-04-29 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Ovarian Neoplasms
Keywords: immunotherapy; monoclonal; antibody; Stage III ovarian epithelial cancer; Stage IV ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — oregovomab

INTERVENTIONS:
Drug: oregovomab

SUMMARY:
In this study, patients will be randomized to one of three dose regimen groups. Each dose of OvaRex MAb-B43.13 is 2 mg by slow intravenous administration.

Group 1 will receive two doses, one month apart.

Group 2 will receive three consecutive monthly doses, then at 12-week intervals through 2 years or until disease relapse up to a total of 9 doses.

Group 3 will receive six consecutive monthly doses, then at 12-week intervals through 2 years or until disease relapse up to a total of 11 doses.

The study will compare the time to disease relapse of patients who demonstrate an immune response to OvaRex MAb-B43.13 with time to disease relapse of those who do not demonstrate an immune response to OvaRex MAb-B43.13. Differences in the percentage of patients demonstrating an immune response in each dose regimen group will also be assessed.

ELIGIBILITY:
Inclusion Criteria

* Histological diagnosis of epithelial adenocarcinoma of ovarian, tubal or peritoneal origin and disease is classified as FIGO Stage III or IV.
* Functional Performance Status < or = 2 by ECOG scale or > or = 60% on Karnofsky scale.
* Medical assessment consistent with prognosis for an expected survival of at least 6 months.
* Serum CA125 level >35 U/mL prior to or at initial surgery. Alternatively, serum CA125 level > or = 100 U/mL and immunohistochemical evidence of tumor tissue expressing CA125.
* Presence of residual disease that is either (a) visible to or palpable by the surgeon at the completion of the staging laparotomy procedure, or (b) microscopic disease remaining following the staging laparotomy procedure.
* Received chemotherapy that included cisplatin or carboplatin following appropriate staging procedure.
* Complete clinical response to primary treatment protocol, which included laparotomy followed by platinum-based adjuvant chemotherapy.

Exclusion Criteria:

* First dose of study medication must be within 10 weeks of completing last dose of primary chemotherapy.
* Not more than one prior regimen of chemotherapy. A change of chemotherapy agents is permitted during the patient's primary therapy provided that the change is considered to be part of the initial chemotherapy treatment regimen.
* No whole abdomen, abdominopelvic or pelvic radiotherapy, surgery or chemotherapy within 4 weeks prior to first dose of study drug.
* No immunotherapy (interferons, tumor necrosis factor, other cytokines or biological response modifiers, or BCG vaccines) within the previous 6 weeks of first study dose. Patients who have received hemopoietic factors are acceptable.
* No previous treatment with murine monoclonal antibodies for diagnostic or therapeutic purposes.
* No compromised hematopoietic function defined as a hemoglobin <8.0 g/dL or lymphocyte count <300 mm3 or neutrophil count <1000 mm3 or platelet count <100,000 mm3.
* No hepatic dysfunction defined as a bilirubin >1.5 times the upper normal limits.
* No severe renal dysfunction defined as serum creatinine >1.6 mg/dL.
* While pregnancy is unlikely in view of the disease and previous surgery, patients who the investigator considers may be at risk of pregnancy will have a pregnancy [beta-HCG] test and will be using a medically approved contraceptive method. Patients who are breast-feeding are also excluded.
* No active autoimmune disease (e.g., rheumatoid arthritis, SLE, ulcerative colitis, Chrohn?s Disease, MS, ankylosing spondylitis).
* No known allergy to murine proteins, or prior documented anaphylactic reaction to any drug.
* Not on chronic treatment with immunosuppressive drugs such as cyclosporin, ACTH, or corticosteroids.
* No active infection causing fever.
* No previous splenectomy.
* No recognized immunodeficiency disease including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia; no acquired, hereditary, or congenital immunodeficiencies.
* No uncontrolled diseases or illness other than this cancer. Patients with chronic diseases that are well controlled (e.g., diabetes mellitus, hypertension) are eligible.
* No significant cardiovascular abnormalities (uncontrolled hypertension, CHF (NYHA Classes II-IV), uncontrolled angina, or uncontrolled arrhythmias).
* No concurrent illness or chronically taking medication that could confound the results of the study, preclude the patient from completing the study or mask an adverse reaction.
* No concurrent malignancy (except non-melanoma of the skin or in situ carcinoma of cervix), unless curative treatment was received and patient has been disease-free for > or = 5 years.
* No other investigational drugs within 30 days of enrollment.
* No contraindications present to the use of pressor agents.
* Inability to read or understand, and/or unwilling to sign a written consent form which must be obtained prior to treatment.
* Only tumors of low malignant potential or with noninvasive disease.
* Not more than one interval debulking procedure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102
Dates: Start 2000-09; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (12):
  - Gynecologic Oncology Associates, Newport Beach, California
  - Stanford University Medical Center, Stanford, California
  - Walt Disney Memorial Cancer Institute, Orlando, Florida
  - St. Joseph's Regional Medical Center, South Bend, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Parker Hill Oncology & Hematology, Boston, Massachusetts
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Baptist Hospital of East Tennessee, Knoxville, Tennessee
  - Texas Oncology, P.A., Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Swedish Medical Center Tumor Institute, Seattle, Washington
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Centre Hospitalier Universitaire de Sherbrooke - Hopital Fleurimont, Fleurimont, Quebec
  - SMBD Jewish General Hospital, Montreal, Quebec